CLINICAL TRIAL: NCT07004439
Title: A Post-market Registry Study Based on Standard Clinical Care to Assess Safety and Performance of RefluxStop™ in the Treatment of Gastroesophageal Reflux Disease (GERD) in General Hospital Practice
Brief Title: A Post-market Registry to Assess Safety and Performance of RefluxStop™ in the Treatment of GERD in General Hospital Practice
Acronym: RESTORE500
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Implantica CE Reflux Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RXI006
Record Dates: First submitted 2025-05-27; First posted 2025-06-04 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-03

CONDITIONS: Gastroesophageal Reflux Disease
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single arm: intervention (Other): Single arm registry: all enrolled patients will be implanted with RefluxStopTM
  Interventions: Device: RefluxStop™ implantation

INTERVENTIONS:
Device: RefluxStop™ implantation — Standard surgical technique for implantation RefluxStop™, as described in the Instructions for Use

SUMMARY:
A post-market retrospective and prospective, open label, multicenter, single-arm registry study using standard clinical procedures to record available and/or new data to evaluate the safety and performance of RefluxStop™ for the treatment of subjects suffering from GERD.

Following surgery, patients will have follow-ups visits at 3 and 6 months and annually up to 7 years.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to provide informed consent and to participate in the registry study;
2. Age ≥ 18 years or according to local legal age of adulthood at the location of the test site if older;
3. Documented GERD present for ≥ 6 months. Typical symptoms are defined as heartburn;
4. 24-hour pH or impedance pH monitoring proven GERD with pH measurement, off PPI therapy for at least 7 days prior to testing. (Total distal esophageal pH must be < 4 for ≥ 4.5% of total time during a 24-hour monitoring) and/or total reflux episodes >55 or weekly acid >26 for > 5 seconds, all measured 5 cm above LES);
5. Suitable to undergo general anaesthesia and is a suitable laparoscopic surgery candidate as determined by the investigator.

Exclusion Criteria:

1. Hiatal Hernia larger than 8 cm;
2. Known presence of delayed gastric emptying, if no other cause for acid reflux could be diagnosed. Patients with substantially weak peristalsis (manometry DCI value 100-200) in esophagus measured during manometry would continue the simplified contrast swallow x-ray to perform a simplified two-hour gastric emptying contrast swallow
3. History of bariatric surgery wherein the stomach fundus has been extirpated;
4. Female subjects who are pregnant;
5. Known sensitivity or allergies to silicone materials;
6. Intraoperative findings determined by the investigator that may result in unfavorable conduct of the registry procedure (as outlined in the IFU);
7. Subjects that are unable to comply with the registry requirements (for example due to major psychiatric disorder or are considered otherwise unsuitable for participation in the clinical investigation according to the investigator's judgement).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2025-09-15 (Estimated); Primary Completion 2029-08-01 (Estimated); Study Completion 2035-08-01 (Estimated)

PRIMARY OUTCOMES:
Reduction of Patient Reported Outcome - Side effects (PROS) | 1 year
  Patient Reported Outcome - Side effects (PROS) combine the established side effects: Dysphagia, Odynophagia, Inability to Belch, Inability to Vomit, and worsened Gas bloating, compared to baseline

SECONDARY OUTCOMES:
Incidence of safety events | 3 and 6 months and years 1 to 7
  Safety events include: SADEs, SAEs, ADEs, procedure-related or unknown AEs and DDs
Reduction of Patient Reported Outcome - Side effects (PROS) | 6 months and years 2 to 7
  Patient Reported Outcome - Side effects (PROS) combine the established side effects: Dysphagia, Odynophagia, Inability to Belch, Inability to Vomit, and worsened Gas bloating, compared to baseline

CONTACTS AND LOCATIONS:
Locations (5):
- Klinikum Friedrichshafen GmbH, Friedrichshafen, Germany
- Spain (4):
  - H. Universitario Getafe, Getafe, Madrid
  - H. La Mancha Centro, Alcázar de San Juan
  - H. Infanta Sofía, Madrid
  - H. Ramón y Cajal, Madrid

IPD SHARING:
Plan to Share IPD: No